CLINICAL TRIAL: NCT03163524
Title: Applying Behavioural Insights to Improve Take up of Sexual and Reproductive Health Services
Brief Title: Behavioural Insights to Improve Take up of SRH Services (Uganda)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marie Stopes International (Other)
Collaborators: Ideas42 (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 007-15
Record Dates: First submitted 2016-07-18; First posted 2017-05-23 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Health Behavior
Keywords: family planning; reproductive health; m-health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (modified text) (Experimental): The treatment group will receive a modified text of the current e-coupon. They will also receive notification that they have been enrolled in the study via a second text. They will also receive a series of text message reminders to redeem their e-coupons at intervals of 6, 13 and 18 days after coupon origination.
  Interventions: Other: e-Coupon Text Modification and Reminders
- Control group (standard text) (Sham Comparator): Participants receive control text (SMS) message, which contains a numeric coupon code and no additional text to the standard coupon.
  Interventions: Other: e-Coupon standard text

INTERVENTIONS:
Other: e-Coupon Text Modification and Reminders — The treatment group will receive a modified text of the current e-coupon. They will also receive notification that they have been enrolled in the study via a second text. They will also receive a series of text message reminders to redeem their e-coupons at intervals of 6, 13 and 18 days after coupon origination.
  Arms: Treatment group (modified text)
Other: e-Coupon standard text — Participants receive control text (SMS) message, which contains a numeric coupon code and no additional text to the standard coupon.
  Arms: Control group (standard text)

SUMMARY:
This is a randomised controlled trial to test the impact of a modified e-coupon service, delivered through SMS, on uptake of sexual and reproductive health services among women calling a free hotline in Uganda.

DETAILED DESCRIPTION:
The overall goal of the proposed research project is to increase uptake of sexual and reproductive health (SRH) services among clients who call into Marie Stopes Uganda's free hotline. The study seeks to achieve this goal by using behavioural economics to design interventions to increase redemptions of e-coupons distributed to hotline clients. The intervention will include modifying the text message sent to e-coupon recipients as well as sending follow-up texts reminding clients to use their coupons. The impact of the intervention will be evaluated using a randomized controlled trial (RCT). The intervention will be implemented and data will be collected regularly over a period of approximately 12 months. Strict confidentiality procedures in line with Marie Stopes International's best practices will be put into place to ensure that information made public or otherwise distributed outside the principle investigators and other key personnel cannot be linked to any individual respondents. Results from the study will be published in a report, among other outputs, and the outcomes will be shared within MSI as well as with the wider SRH community.

ELIGIBILITY:
Inclusion Criteria:

* Callers to the call centre who are over the age of 18, receive an e-coupon, and consent to participate in the research.

Exclusion Criteria:

* Callers who are below the age of 18, non-recipients of e-coupons, and those who receive e-coupons but do not consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Increase in e-coupon redemption in MSU centres | 6 months
  Increase in proportion of e-coupons redemmed in MSU centres within 6 months of intervention
Increase in SRH service uptake in MSU centres | 6 months
  Increase in the proportion of participants taking up an SRH service (of any kind) in an MSU centre within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Aujo, Principal Investigator — Marie Stopes International; Andrew Fertig, PhD, Principal Investigator — Ideas42; Karina Lorenzana, Principal Investigator — Ideas42; Andrew Gidudu, MSc, Principal Investigator — Marie Stopes International
Locations (1):
- Marie Stopes Uganda call centre, Kampala, Uganda